CLINICAL TRIAL: NCT06152471
Title: A Randomized Double-blind Placebo Controlled Phase 3 Trial on the Effect of Salovum™ and SPC-Flakes™ on Abemaciclib-induced Gastrointestinal Toxicity in Early Breast Cancer - the ASF-BC Study
Brief Title: Effect of Salovum™ and SPC-Flakes™ on Abemaciclib-induced Gastrointestinal Toxicity in Early Breast Cancer
Acronym: ASF-BC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henrik Lindman (Other)
Responsible Party: Sponsor-Investigator, Henrik Lindman, Coordinating Investigator, Uppsala University Hospital
Organization: Uppsala University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Version 1.3, 30May2022
Record Dates: First submitted 2023-10-19; First posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Early-stage Breast Cancer; Diarrhea; Adverse Drug Event
Keywords: Early Breast cancer; Abemaciclib induced diarrea
MeSH Terms: conditions — Breast Neoplasms; Diarrhea; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Intervention Model Description: Randomization 1:1 to investigational product or placebo
Who Masked: Participant, Investigator
Masking Description: double-blind, placebo controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Salovum egg powder high in antisecretory factor, 4 g/sachet. Four sachets, ie 16 gr q 8 hours for 6 days before start of abemaciclib
  SPC-flakes flat dose 75gr/day in parallel and during first 12 weeks of treatment with abemaciclib
  Interventions: Drug: SPC-flakes; Drug: Salovum
- Placebo Comparator (Placebo Comparator): Placebo, identical to investigational product but without antisecretory factor.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPC-flakes — Aktive drug
  Arms: Experimental
Drug: Salovum — Active drug
  Arms: Experimental
Drug: Placebo — Placebo drugs
  Arms: Placebo Comparator

SUMMARY:
The present study aims to investigate a proactive strategy including Salovum™ and SPC-flakes to prevent the occurrence of abemaciclib-induced diarrhea in patients with early breast cancer.

DETAILED DESCRIPTION:
In patients with high-risk luminal breast cancer, the addition of CDK 4/6-inhibitor abemaciclib to adjuvant endocrine therapy for two years has been associated with improved disease-free survival and is now recommended from national and international guidelines as the preferred treatment strategy for this patient group. However, patients treated with abemaciclib have higher risk of diarrhea which primarily occurs during the first three months from treatment initiation and seems to impact patients' quality of life. As a result, early and proactive strategies to reduce the occurrence of diarrhea from the initiation of abemaciclib should be investigated to ensure that patients in whom adjuvant abemaciclib is recommended can complete their treatment as planned.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Histologically confirmed diagnosis of luminal breast cancer.
* No clinical evidence of metastatic disease.
* Planned to start abemaciclib in adjuvant setting (according to current national guidelines).
* Signed informed consent.

Exclusion Criteria:

* Contraindications to the investigational product, e g known or suspected hypersensitivity to the investigational products or expected inability to their use in accordance with the protocol.
* Lack of suitability for participation in the study, e g expected difficulties to follow the protocol procedures, as judged by the investigator.
* Prior exposure to abemaciclib.
* Prior exposure to Salovum or SPC-flakes.
* Past or present history of inflammatory bowel disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-06-07 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Abemaciclib induced diarrhea - STIDAT | Three months
  ● Occurrence of any-grade (mild, moderate, severe) diarrhea according to the Systemic Treatment-Induced Diarrhea Assessment Tool (STIDAT; patient-reported outcome).

SECONDARY OUTCOMES:
Occurrence of abemaciclib induced diarrhea - CTCAE | Three months
  Occurrence of any-grade diarrhea according to CTCAE v. 5.0
QoL using FACT-B | Three months
  The tool is FACT-B
QoL using FACT-GP5 | Three months
  The tool is FACT-GP5
QoL using FACIT-D | Three months
  The tool is FACIT-D
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] besides diarrhea. | Three months
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0, besides diarrhea.
Rate of patients that stop or interrupt treatment with investigational products | Three months
  Rate of patients that stop or interrupt treatment with Salovum and SPC-flakes/placebo during planned study time.
Rate of patients that stop or interrupt treatment with abemaciclib | Two years
  Rate of patients that stop or interrupt treatment with abemaciclib during the planned treatment time of two years.
Sick leave | Two years
  Sick leave duration
Breast cancer recurrence | Two years
  Breast cancer recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Lindman, MD, PhD, Principal Investigator — Uppsala University Hospital
Locations (7):
- Sweden (7):
  - General Hospital of Eskilstuna, Eskilstuna
  - General Hospital of Falun, Falun
  - General Hospital of Gävle, Gävle
  - University Hospital Örebro, Örebro
  - General Hospital, Sundsvall
  - Uppsala University Hospital, Uppsala
  - General Hospital Västerås, Västerås